CLINICAL TRIAL: NCT07074886
Title: A Phase II, Randomized, Open-label, Parallel Group, Multicenter Study to Assess Bioequivalence of Two Subcutaneous Formulations of Ocrelizumab in Patients With Multiple Sclerosis
Brief Title: A Study to Assess Bioequivalence of Two Subcutaneous (SC) Formulations of Ocrelizumab in Participants With Multiple Sclerosis (MS)
Acronym: PORTAMENTO
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CN45320; 2024-517980-22-00 (EU CTIS Number)
Record Dates: First submitted 2025-07-17; First posted 2025-07-20 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ocrelizumab Test Formulation (Experimental): Participants will receive ocrelizumab test formulation, as SC injection, as per a pre-defined dosing regimen during the controlled phase and continuation phase.
  Interventions: Drug: Ocrelizumab Test Formulation
- Ocrelizumab Reference Formulation (Active Comparator): Participants will receive ocrelizumab reference formulation, 920 mg, as SC injection, on Day 1 during the controlled phase. Thereafter, participants will receive ocrelizumab test formulation, as SC injection, as per a pre-defined dosing regimen during the continuation phase.
  Interventions: Drug: Ocrelizumab Test Formulation; Drug: Ocrelizumab Reference Formulation

INTERVENTIONS:
Drug: Ocrelizumab Test Formulation — Ocrelizumab test formulation will be administered as per the schedule specified in the respective arm.
  Other Names: RO4964913
Drug: Ocrelizumab Reference Formulation — Ocrelizumab reference formulation will be administered as per the schedule specified in the respective arm.
  Other Names: RO4964913
  Arms: Ocrelizumab Reference Formulation

SUMMARY:
The main purpose of this study is to assess the bioequivalence of ocrelizumab SC test formulation to the marketed ocrelizumab SC reference formulation in participants with either relapsing multiple sclerosis (RMS) or primary progressive multiple sclerosis (PPMS). The study consists of 2 phases: a controlled phase, where participants in each group will receive one dose of test or reference formulation and a continuation phase, where all participants in both groups will receive ocrelizumab SC test formulation.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of RMS or PPMS according to the revised McDonald 2017 criteria (Thompson et al. 2018) or the most current McDonald criteria at the time of study start
* Expanded Disability Status Scale (EDSS) score, 0-6.5, inclusive, at screening

Exclusion Criteria:

* Participants who have previously received anti-cluster of differentiation (CD) 20s (including ocrelizumab) less than 2 years before screening
* Participants who have previously received anti-CD20s (including ocrelizumab) more than 2 years before screening if one of the following conditions is met: B-cell count is below lower limit of normal (LLN), or the discontinuation of the treatment was due to safety reasons
* History of confirmed or suspected progressive multifocal leukoencephalopathy (PML)
* History of cancer, including hematologic malignancy and solid tumors, within 10 years of screening
* Immunocompromised state
* Sensitivity or intolerance to any ingredient (including excipients) of ocrelizumab
* History of severe allergic or anaphylactic reactions to humanized or murine monoclonal antibodies
* Any concomitant disease that may require chronic treatment with systemic corticosteroids or immunosuppressants during the course of the study
* Significant, uncontrolled disease, such as cardiovascular, pulmonary, renal, hepatic, endocrine or gastrointestinal, or any other significant disease that may preclude participation in the study
* Lack of peripheral venous access
* Previous treatment with cladribine, atacicept, and alemtuzumab
* Any previous treatment with bone marrow transplantation and hematopoietic stem cell transplantation
* Any previous history of transplantation or anti-rejection therapy
* Positive screening tests for active, latent, or inadequately treated hepatitis B virus (HBV)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Estimated)
Dates: Start 2025-11-13 (Actual); Primary Completion 2027-01-31 (Estimated); Study Completion 2030-10-30 (Estimated)

PRIMARY OUTCOMES:
Area Under the Serum Concentration-time Curve Over the First 12 Weeks Post-dose (AUC0-12W) of Ocrelizumab | Up to 12 weeks
Maximum Serum Concentration (Cmax) of Ocrelizumab | Up to 12 weeks

SECONDARY OUTCOMES:
Number of Participants With Adverse Events (AEs) | Up to 168 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (41):
- United States (4):
  - Profound Research, LLC, Carlsbad, California
  - Advanced Neurology of Colorado, LLC, Fort Collins, Colorado
  - Neurology Associates PA, Maitland, Florida
  - Hope Neurology, Knoxville, Tennessee
- Argentina (6):
  - Centro de Especialidades Neurológicas y Rehabilitación - CENyR, CABA, Buenos Aires
  - Focus CECIC, CABA, CABA / Buenos Aires
  - INECO Neurociencias Orono, Rosario, Santa Fe Province
  - IME - Instituto Médico Especializado, Buenos Aires
  - Centro de Investigacion en Enfermedades Reumaticas CIER, Ciudad Autonoma Buenos Aires
  - Sanatorio del Sur S.A., San Miguel de Tucumán
- Brazil (8):
  - Santa Casa de Misericordia de Salvador, Salvador, Estado de Bahia
  - Freire Pesquisa Clinica, Belo Horizonte, Minas Gerais
  - Instituto de Neurologia de Curitiba, Curitiba, Paraná
  - Cpn - Centro de Pesquisa Neurologica Porto Alegre Ltda, Porto Alegre, Rio Grande do Sul
  - Núcleo de Pesquisa do Rio Grande do Sul, Porto Alegre, Rio Grande do Sul
  - Instituto do Cerebro do Rio Grande do Sul, Porto Alegre, Rio Grande do Sul
  - Clinica Neurológica e Neurocirúrgica de Joinville, Joinville, Santa Catarina
  - Centro de Pesquisas Clinicas - CPCLIN, São Paulo, São Paulo
- Charite - Universitätsmedizin Berlin, Berlin, Germany
- Italy (4):
  - AO.U. Policlinico Riuniti Foggia, Foggia, Apulia
  - Policlinico Tor Vergata Dip. Neuroscienze-Clinica Neurologica-UOSD Sclerosi Multipla, Rome, Lazio
  - NCL Institute Neuroscience, Rome, Lazio
  - IRCCS Istituto Neurologico Neuromed, Pozzilli, Molise
- Mexico (4):
  - Clinstile S.A de C.V., Mexico City, Mexico CITY (federal District)
  - Inovacion y Desarrollo en ciencias de la salud, Mexico City, Mexico CITY (federal District)
  - Neurociencias Prisma, A.C, San Luis Potosí City, San Luis Potosí
  - Neurociencias Estudios Clinicos S.C., Culiacán, Sinaloa
- Poland (6):
  - ProNeuro Centrum Medyczne, ?ory
  - Neurocentrum Bydgoszcz sp z o.o, Bydgoszcz
  - Centrum Neurologii Krzysztof Selmaj, Lodz
  - Instytut Zdrowia Dr Boczarska-Jedynak Sp. z o.o. Sp. k., Oświęcim
  - Nmedis sp. z o.o., Rzeszów
  - IBISMED Wielospecjalistyczne Centrum Medyczne, Zabrze
- Spain (8):
  - Hospital de Gran Canaria Dr. Negrín, Las Palmas de Gran Canaria, LAS Palmas
  - Hospital Universitario Virgen de Arrixaca, EL Palmar (EL Palmar), Murcia
  - Complejo Hospitalario Universitario de Albacete, Albacete
  - Hospital General Universitario de Alicante, Alicante
  - Hospital Universitari Vall dHebron (CEMCAT), Barcelona
  - Hospital Universitario de la Princesa, Madrid
  - Hospital Ramon y Cajal, Madrid
  - Hospital Universitario Virgen Macarena, Seville

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing